CLINICAL TRIAL: NCT03533075
Title: A Pilot Effectiveness Trial of the Teachable Moment Brief Intervention (TMBI) for Veterans Hospitalized Following a Suicide Attempt
Brief Title: Teachable Moment Brief Intervention for Veterans Following a Suicide Attempt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisville VA Medical Center (U.S. Federal Agency)
Collaborators: University of Louisville (Other)
Responsible Party: Principal Investigator, Stephen O'Connor, Ph.D., Research Facilitator, Louisville VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00466
Record Dates: First submitted 2018-04-26; First posted 2018-05-22 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Suicide, Attempted
MeSH Terms: conditions — Suicide, Attempted

STUDY DESIGN:
Intervention Model Description: Participants will be assigned in even numbers to TMBI + follow-up consultation or care as usual.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will remain blinded to the treatment condition for all participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teachable Moment Brief Intervention (Experimental): The TMBI is informed by evidence based strategies to collaboratively identify 1) drivers of suicidal ideation, 2) functional aspects of the recent suicide attempt, 3) the patient's relationship with the concept of suicide, 4) what has been lost and gained as a result of the suicide attempt, 5) short term management suicide prevention management strategies, and 6) documentation of factors to address in a suicide-specific treatment plan.
  Interventions: Behavioral: Teachable Moment Brief Intervention
- Care as Usual (No Intervention): Usual care at Veterans Affairs Medical Centers (VAMC) for Veterans who have attempted suicide involves psychiatric evaluation/treatment and ongoing medical stabilization.

INTERVENTIONS:
Behavioral: Teachable Moment Brief Intervention — Behavioral intervention informed by Collaborative Assessment and Management of Suicidality and Dialectical Behavior Therapy/Cognitive Behavior Therapy to assist in positive recovery trajectory following a suicide attempt
  Arms: Teachable Moment Brief Intervention

SUMMARY:
The overall objective is to determine the acceptability and feasibility of the Teachable Moment Brief Intervention (TMBI) + follow-up consultation for Veterans treated on an inpatient psychiatry unit following a suicide attempt. The study will also determine whether there is a signal of effectiveness supporting the TMBI in improving the recovery trajectory of Veterans following discharge to the community.

DETAILED DESCRIPTION:
A total of 50 patients will be recruited from the inpatient psychiatry unit for the study. A member from the research team will obtain informed consent for the participants and then administer the baseline assessment battery. Patients will then be randomized to either (a) an experimental group receiving TMBI + follow-up consultation or (b) a group receiving care as usual. Patients randomized to the experimental group will receive the intervention prior to discharge from the hospital, most likely on the same day as the baseline assessment battery. Patients receiving the experimental intervention will then be asked to complete a brief post-intervention client satisfaction survey administered by a research team member. All study participants will then complete telephone follow-up assessments at 1 and 3-month time points administered by members of the research team and supervised by the PI. Additionally, patient electronic medical records will be abstracted to document the following health services and clinical characteristics in the 12 months following enrollment in the study: death for any reason, inpatient hospitalization (both medical/surgical and psychiatric), emergency department visits, suicide attempt and other forms of self-directed violence, all outpatient appointments with VA service providers, and diagnosis. The PI will rate the TMBI sessions for the interventionists. When the PI delivers the intervention, a trained member of the research team will review the PI's sessions and rate for adherence. The intervention will consist of no more than 90 minutes (expected mean is 45 minutes for the intervention based upon previous studies of the TMBI) of 1:1 interaction with a study clinician. The baseline assessment battery will take approximately 30 minutes, the post-intervention measure will take approximately 5 minutes, and the 1 and 3-month assessment batteries will take approximately 30 minutes. The PI and potentially 2 to 3 members of the Suicide Prevention Program will provide the intervention to ~25 randomized patients.

Notes will be kept on patients who decided to drop out of the intervention and/or the study. We will examine the mean and standard deviation for the total score and individual items on the Client Satisfaction Questionnaire. Notes will be kept documenting all contacts for recruitment and the number of eligible patients per month. Reasons for inclusion and exclusion of potential participants will be documented as well as reasons participants give for choosing not to participate. Number of patients enrolled and randomized each month will be documented. Notes will be kept of rates of on-time outcome assessments and days late and any assessments missed or participants lost to contact.

Descriptive statistics for demographic and clinical variables will be tabulated. All scales will be scored and subscales described. This process will include examining the data for missing values, appropriate ranges, and outliers. Although the randomization design should ensure balance between the two groups, it is essential to control for any known confounders in the design and analysis to prevent a biased assessment of the brief intervention effect. Any baseline demographic or clinical variables found to be statistically significant in the analysis will be included as covariates in all analytic models. We will use an intent-to-treat sample to complete our analyses. We will utilize mixed-effects regression models to obtain between-groups effect sizes for the impact of the TMBI + consultation on elevating motivation, hope, reasons for living and social connection.

ELIGIBILITY:
Inclusion Criteria:

1. Veteran service member
2. Recently admitted to an inpatient psychiatry unit at the VAMC site following a suicide attempt
3. 18 or more years of age
4. Consents to participate in baseline and follow-up interviews and gives permission to review records for previous year and subsequent year.
5. Consents to randomization and participation in TMBI + follow-up or Care as Usual
6. Consents to audio recording in order for PI to conduct adherence rating

Exclusion Criteria:

1. Significant psychosis, cognitive, or other problems that prevent participant from understanding the study procedures or renders them unable to provide informed consent (suggesting that psychosocial therapeutic care is contra-indicated)
2. Judicially-ordered to treatment (e.g., subsequent to domestic violence) such that participation in study procedures could not be considered voluntary and participant is not free to drop out without significant negative consequences.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Changes in Stages of Change Questionnaire, which measures motivation | 3 months
  18-item measure that measures motivation to engage in treatment/work on problems. Total score will be summed from all items, with range from 18 (low motivation) to 90 (high motivation). Four subscales will also be reported as follows: Precontemplation ranges from 5 (low) to 25 (high) with higher scores indicating higher motivation. Contemplation ranges from 4 (low) to 20 (high) with higher scores indicating higher motivation. Action ranges from 5 (low) to 25 (high) with higher scores indicating higher motivation. Maintenance ranges from 4 (low) to 20 (high) with higher scores indicating higher motivation.
Changes in Reasons for Living Inventory | 3 months
  48-item measure that rates the importance of different reasons why people choose not to kill themselves. Total score will be reported, which ranges from 48 (low reasons for living) to 288 (High reasons for living).
Changes in State Hope Scale | 3 months
  6-item measure of ongoing self-directed thinking. Total score will be reported, which ranges from 6 (low hope) to 48 (high hope).
Changes in Interpersonal Needs Questionnaire, which measures constructs of thwarted belongingness and perceived burdensomeness. | 3 months
  15-item measure of the extent to which individuals feel connected to others (i.e., belongingness) and like a burden on people in their lives (i.e., perceived burdensomeness). Subscale total scores for thwarted belongingness and perceived burdensomeness will be reported. For thwarted belongingness, scores range from 9 (low) to 63 (high). For perceived burdensomeness, scores range from 6 (low) to 42 (high).
Changes in Beck Scale for Suicide Ideation | 3 months
  19-item assessment used to evaluate the current intensity of the patient's specific attitudes toward, behavior, and plans to commit suicide. Total score will be reported which ranges from 0 (no suicidal ideation) to 38 (high suicidal ideation)
Suicide Attempt Self-Injury Count | 3 months
  two-page instrument determining for the first, most recent, and most severe suicide attempt or non-suicidal self-injury (SASI) the date, method of SASI attempt used in index and previous attempts according to the definitions of Linehan et al. (e.g., using definitions of self-inflicted injuries which include situations of actual tissue damage and situations where tissue damage would have occurred except for outside intervention or sheer luck [e.g., firearm jammed]), intent to die (i.e., intent to die, ambivalent, no intent to die), highest level of medical treatment received, and lethality

SECONDARY OUTCOMES:
Outpatient Health Services Engagement | 12 months
  all outpatient appointments with VA service providers using electronic health record data
Acute Care Health Services | 12 months
  inpatient hospitalization (both medical/surgical and psychiatric) and emergency department visits using electronic health record data
Self-Directed Violence | 12 months
  All documented self-directed violence across 12 months using electronic health record data

CONTACTS AND LOCATIONS:
Overall Officials: Stephen O'Connor, PhD, Principal Investigator — Robley Rex VA Medical Center
Locations (1):
- Robley Rex VA Medical Center, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617